CLINICAL TRIAL: NCT01915420
Title: Postmarketing Surveillance Registry to Monitor Everolimus-eluting Bioresorbable Vascular Scaffold Following Rotational Atherectomy for the Treatment of Complex Coronary Lesions - The ASSURE ROT Registry
Brief Title: The ASSURE ROT Registry: Bioresorbable Vascular Scaffold Following Rotablation for Complex Coronary Lesions
Acronym: ASSURE ROT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical Care Center Prof. Mathey, Prof. Schofer, Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: ASSURE ROT
Record Dates: First submitted 2013-07-29; First posted 2013-08-02 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Cardiovascular Diseases; Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Coronary Restenosis; Heart Diseases; Coronary Stenosis; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases
Keywords: Drug eluting stent; Bioabsorbable; Bioresorbable; Coronary Stent; Scaffold; Stents; Angioplasty; Coronary Artery Disease; Stentthrombosis; Rotational atherectomy
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Coronary Restenosis; Heart Diseases; Coronary Stenosis; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The registry aims to evaluate the safety, performance and efficacy of the Everolimus-eluting bioresorbable vascular scaffold (BVS) system following rotational atherectomy in patients with complex de novo native coronary artery lesions in all-day clinical practice.

DETAILED DESCRIPTION:
Bioresorbable scaffolds are transient implants. They act like drug-eluting metallic stents (DES) during the first 3 months by supporting the vessel wall thereby keeping the artery patent. Subsequently, resorption of the scaffold begins and its structure loosens. As a result of everolimus release, neointimal growth is inhibited similar to DES. Finally the implant is reabsorbed completely in about 2-3 years. BVS in terms of late stent thrombosis may be safer than DES. Transiently scaffolded vessels may regain their natural curvature and angulation as well as response to nitroglycerine and endothelial function.

ELIGIBILITY:
The recommendation to implant BVS in an individual patient in whom rotational atherectomy of a complex target lesion has been conducted, is purely based on clinical grounds. These are determined by the instructions for use (IFU) of the BVS and by the clinical experience accumulated so far from clinical studies.These studies suggest that the BVS should be implanted under certain conditions, which are determined by the patient and the coronary lesion treated:

Eligible:

Regarding to patient

* Patient ≥ 18 and ≤ 75 years with a live expectancy of at least 5 years with ischemic heart disease (chronic, NSTEMI and unstable angina) due to one or more complex de novo native coronary artery lesions
* Patients with evidence of myocardial ischemia

Regarding to lesion

* Reference vessel diameter ≥ 2.5 mm and ≤ 3.8 mm, visually estimated or by online QCA
* Percent diameter stenosis ≥ 50% and < 100%, visually estimated or by online QCA
* TIMI ≥1
* Previous interventions of target vessel lesions should have been done ≥ 6 months prior to index procedure and > 10 mm distal to the target lesion
* Previous interventions of non-target vessel lesions should have been done ≥ 30 days prior to index procedure

Not eligible:

Regarding to patient

* Patient in whom antiplatelet therapy and/or anticoagulant therapy is contraindicated
* Patient with a known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, clopidogrel, ticlopidine, prasugrel and ticagrelor, everolimus, poly (L-lactide), poly (D,L-lactide), or platinum, or with contrast sensitivity, who cannot be adequately premedicated
* Patient has a known diagnosis of acute myocardial infarction (STEMI) within 72 hours preceding the index procedure and CK and CK-MB have not returned within normal limits at the time of procedure
* Patient is currently experiencing clinical symptoms consistent with STEMI
* Patient has current unstable arrhythmias
* Patient has a known left ventricular ejection fraction < 30%
* Patient has received a heart transplant or any other organ transplant or is waiting for any organ transplant
* Patient receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or after procedure
* Patient is receiving immunosuppression therapy and has known immunosuppressive or autoimmune disease
* Patient is receiving or scheduled to receive chronic anticoagulation therapy
* Elective surgery is planned within the first 6 month after the procedure that will require discontinuing either aspirin or clopidogrel
* Patient has a platelet count < 100 000 cells/mm3 or > 700 000 cells/mm3, a WBC of
* < 3000 cells/mm3, or documented or suspected liver disease
* Patient has known renal insufficiency
* Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Patient has cerebrovascular accident or transient ischemic neurological attack within the past six month
* Patient has had a significant GI or urinary bleed within the past six months
* Patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion
* Patient has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause noncompliance with the clinical study plan, confound the data interpretation or is associated with a limited life expectancy (i.e., les than one year)
* Women of childbearing potential who have not undergone surgical sterilization or are not post- menopausal

Regarding to lesion

Target lesion(s) meets none of the following criteria:

* Aorto-ostial location
* Left main location
* Located within 2 mm of the origin of LAD or LCX
* Located within an arterial or saphenous vein graft or distal to a diseased (defined as vessel irregularity per angiogram and > 20% stenosed lesion by visual estimation) arterial or saphenous vein graft
* Ostial lesion > 40% stenosed by visual estimation or side branch requiring predilation
* Excessive tortuosity proximal to or within the lesion (extreme angulation proximal to or within the lesion)
* Restenotic from previous intervention

Target vessel is not containing thrombus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with complex coronary artery lesions
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Event (MACE) | at 24 months
  Composite of ischemia driven target lesion revascularisation (TLR), myocardial infarction and cardiac death

SECONDARY OUTCOMES:
Acute procedural success | At the end of hospital stay (maximum of 7 days)
  Achievement of final in-scaffold residual stenosis of < 50% and TIMI flow 3 of the target site. Successful delivery and deployment of at least one study scaffold at the intended target lesion and successful withdrawal of the delivery system for all target lesions without occurrence of cardiac death, target vessel MI or repeat TLR during hospital stay (maximum of 7 days). In dual target lesion setting both lesions must meet clinical procedure success criteria.
Acute device success | At time of intervention
  Successful delivery and deployment of the first scaffold at the intended target lesion (in overlapping setting both planned scaffolds) and successful withdrawal of delivery system. Attainment of < 50 % residual stenosis and TIMI flow 3 of the target site, using the BVS without the need for other non- study stents.
Scaffold thrombosis | At time of intervention, and at 6, 12, 24, and 36 months
Cardiac death | At time of intervention, and at 6, 12,24, and 36 months
Myocardial infarction | At time of intervention, and at 6, 12, 24, and 36 months
Ischemia driven target lesion revascularisation (TLR) | At time of intervention, participants will be followed for the duration of hospital stay (an expected average of 3 days), at 6, 12, 24, and 36 months
  Composite of ischemia driven target lesion revascularisation (TLR), myocardial infarction and cardial death
Ischemia driven target vessel revascularisation (TVR) | at 6, 12, 24, and 36 month
In-lesion % diameter stenosis | Baseline and final at time of intervention and at 24 months FU
  QCA: Independent CoreLab
Minimal lumen diameter (MLD) | Baseline and final at time of intervention and at 24 months FU
  QCA: Independent CoreLab
In-scaffold late lumen loss (LLL) | At 24 months FU

CONTACTS AND LOCATIONS:
Overall Officials: Detlef G Mathey, Prof. Dr., Principal Investigator — Medical Care Center Prof. Mathey, Prof. Schofer GmbH
Locations (1):
- Medical Care Center Prof. Mathey, Prof. Schofer GmbH, Hamburg, Hamburg, Germany

REFERENCES:
- [Background] Serruys PW, Onuma Y, Dudek D, Smits PC, Koolen J, Chevalier B, de Bruyne B, Thuesen L, McClean D, van Geuns RJ, Windecker S, Whitbourn R, Meredith I, Dorange C, Veldhof S, Hebert KM, Sudhir K, Garcia-Garcia HM, Ormiston JA. Evaluation of the second generation of a bioresorbable everolimus-eluting vascular scaffold for the treatment of de novo coronary artery stenosis: 12-month clinical and imaging outcomes. J Am Coll Cardiol. 2011 Oct 4;58(15):1578-88. doi: 10.1016/j.jacc.2011.05.050. PMID 21958884
- [Background] Dudek D, Onuma Y, Ormiston JA, Thuesen L, Miquel-Hebert K, Serruys PW. Four-year clinical follow-up of the ABSORB everolimus-eluting bioresorbable vascular scaffold in patients with de novo coronary artery disease: the ABSORB trial. EuroIntervention. 2012 Jan;7(9):1060-1. doi: 10.4244/EIJV7I9A168. PMID 21959320
- [Background] Basavarajaiah S, Naganuma T, Latib A, Colombo A. Can bioabsorbable scaffolds be used in calcified lesions? Catheter Cardiovasc Interv. 2014 Jul 1;84(1):48-52. doi: 10.1002/ccd.24939. Epub 2013 Aug 31. PMID 23592566
- [Background] Patel N, Banning AP. Bioabsorbable scaffolds for the treatment of obstructive coronary artery disease: the next revolution in coronary intervention? Heart. 2013 Sep;99(17):1236-43. doi: 10.1136/heartjnl-2012-303346. Epub 2013 Mar 8. PMID 23474621